CLINICAL TRIAL: NCT06183723
Title: Feasible Program of Sustainable Medical Care for People Living With HIV Who Are Difficult to Treat or Marginalized in Taiwan
Brief Title: Optimizing Care for Challenging People Living With HIV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chun-Yuan Lee, MD, Assistant professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-SV(I)-20230081
Record Dates: First submitted 2023-12-06; First posted 2023-12-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Adherence, Medication; HIV Infections; Social Media
Keywords: HIV; Adherence; Social media platform
MeSH Terms: conditions — Medication Adherence; HIV Infections | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- People living with HIV with poor adherence to HAART (Experimental): People living with HIV (PLWH) with adherence below the specific proportion of days covered (PDC), which is defined as the specific level that corresponds to 90% at viral suppression (< 200 copies/mL).
  Interventions: Other: Combination of social-behavior model and eHealth

INTERVENTIONS:
Other: Combination of social-behavior model and eHealth — The study examines how an intervention combining the social-behavior model and eHealth can improve medication adherence among individuals who struggle to follow their medical regimens. The platform offers multiple features including health education, medication reminders, online consultations, chat rooms, news, and Q&A services.
  The intervention and follow-up are based on a 28-day month. The first intervention period runs from the first to the third month post-enrollment, with the introduction of the main features and sharing of health education videos and monthly short films. A follow-up assessment and questionnaire are completed after the third month.
  The second intervention period is between the fourth and sixth months and includes similar features, and face-to-face counseling. New health education videos and monthly short films are shared as well. After the sixth month, another assessment is conducted to evaluate the post-intervention effects.

SUMMARY:
Conduct an intervention combining social and behavioral health models with digital health technologies to improve their adherence to their medication schedules. The success of the intervention is assessed by comparing adherence rates before and after its implementation to see if there's a notable enhancement in how well patients follow their antiretroviral therapy.

DETAILED DESCRIPTION:
This is an intervention strategy for HIV-infected individuals based on their viral load measurements and medication adherence rates, measured by the proportion of days covered (PDC) for the past 365 days. A specific PDC threshold identifies individuals with less than 90% viral suppression at under 200 copies/mL. An intervention approach integrating social and behavioral models with electronic health (eHealth) technology is implemented for cases with a PDC below this threshold. The intervention aims to enhance the patient's adherence to their medication regimen. The effectiveness of this intervention is evaluated by comparing indicators before and after its application to determine if there are significant improvements in the participants' compliance with their antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. PLWH with adherence below the specific proportion of days covered (PDC), which is defined as the specific level that corresponds to 90% at viral suppression (< 200 copies/mL).

Exclusion Criteria:

1. Under 18 years of age.
2. Illiterate.
3. Non-consenting individuals.
4. Less than 365 days from the initial use of antiretroviral drugs to the assessment for inclusion in the study.
5. Inability to obtain complete medication records for the 365 days prior to inclusion.
6. Lack of a smart phone.
7. No willingness to return for follow-up at the participating hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HIV Viral Load from Baseline to 1st and 2nd Follow-Up | At baseline, 84th (+-14) day after enrollment, and 168th (+-14) day after enrollment
  Comparison of HIV viral load (copies/mL) at baseline, 1st follow-up, and 2nd follow-up. The data will be reported as the mean change in viral load from baseline at each time point
Change in CD4 Count from Baseline to 1st and 2nd Follow-Up | At baseline, 84th (+-14) day after enrollment, and 168th (+-14) day after enrollment
  Comparison of CD4 cell count (cells/μL) at baseline, 1st follow-up, and 2nd follow-up. The data will be reported as the mean change in CD4 count from baseline at each time point
Change in Quality of Life Score (WHOQOL-BREF Taiwan Version) from Baseline to 1st and 2nd Follow-Up | At baseline, 84th (+-14) day after enrollment, and 168th (+-14) day after enrollment
  Assessment of participants' quality of life using the WHOQOL-BREF (Taiwan Version) questionnaire at baseline, 1st follow-up, and 2nd follow-up. The results will be reported as the mean score change from baseline at each time point
Change in HIV symptoms index (HIV-SI) in score from Baseline to 1st and 2nd Follow-Up | At baseline, 84th (+-14) day after enrollment, and 168th (+-14) day after enrollment
  Assessment of symptoms using the HIV symptoms index (HIV-SI) at baseline, 1st follow-up, and 2nd follow-up. The results will be reported as the mean score change from baseline at each time point
Change in Self-Reported Antiretroviral Therapy (ART) Medication Adherence from Baseline to 1st and 2nd Follow-Up | At baseline, 84th (+-14) day after enrollment, and 168th (+-14) day after enrollment
  Assessment of self-reported ART medication adherence at baseline, 1st follow-up, and 2nd follow-up. The results will be reported as the proportion of participants who were adherent at each time point, as well as the mean adherence score change from baseline

SECONDARY OUTCOMES:
Change in Proportion of Days Covered (PDC) over the Past 180 Days from Baseline to 1st and 2nd Follow-Up | At baseline and 168th (+-14) day after enrollment
  Assessment of Proportion of Days Covered (PDC) over the Past 180 Days at baseline and 2nd follow-up. The results will be reported as the percentage at each time point, as well as the mean percentage change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yuan Lee, M.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan